CLINICAL TRIAL: NCT01844050
Title: Traditional Chinese Medicine in Individualized Treatment of Patients With Diabetes Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Collaborators: Longhua Hospital (Other); Shanghai Putuo District Center Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 06DZ19728-2; S06DZ19728 (Other: Shanghai University of TCM)
Record Dates: First submitted 2013-04-22; First posted 2013-05-01 (Estimated); Last update posted 2019-06-12 (Actual); Status verified 2013-05

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Chinese herbal medicine; diabetes symptoms
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chinese herbal medicine (Experimental): Individualized Treatment with Chinese herbal
  Interventions: Drug: Chinese herbal medicine
- Placebo (Placebo Comparator): Individualized Treatment with placebo Chinese herbal which Containing 2% of Chinese herbal medicine.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Chinese herbal medicine — According to the traditional Chinese medicine syndrome of subject to make up a prescription within the 35 kinds of chosen Chinese herbal medicine, and the dosage without limitation.
  Arms: Chinese herbal medicine
Drug: Placebo
  Arms: Placebo

SUMMARY:
Based on the Individualized treatment of diabetes symptoms to evaluate the method of syndrome differentiation treatment of Traditional Chinese medicine.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed type 2 diabetes poorly controlled by diet and exercise therapy, and must with any of diabetes symptoms.
* After the diet and exercise therapy, 7.0mmol/l≤FPG≤11.1mmol/l or 8.0mmol/l<2h PG<16mmol/l
* Any type of TCM syndrome, but can be performed within the chosen Chinese herbal medicine.
* Subject is willing to participate and capable of giving informed consent.

Exclusion Criteria:

* Those patients used any drugs for treatment of diabetes within one month.
* Patients with any severe complications of cardiac, cerebric, vascular, hepatic, renal, blood system.
* Patients suffer from acute metabolic disorder including diabetic ketoacidosis or hyperosmotic non-ketotic coma within one month.
* Women who were pregnant, lactating or planned pregnant.
* Allergic constitution and has a history of drug allergy.
* Combined with severe acute or chronic infections.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2008-09; Primary Completion 2009-09 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Total score of diabetes symptoms at 4 weeks | 0 weeks(baseline), 2 weeks, 4 weeks

SECONDARY OUTCOMES:
Change from Baseline Fasting Blood Glucose at 4 weeks | 0 weeks(baseline), 2 weeks, 4 weeks
Change from Baseline blood glucose at 2 hours after meal at 4 weeks | 0 weeks(baseline), 2 weeks, 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kaixian Chen, Ph.D, Study Chair — Shanghai Universitu of TCM
Locations (1):
- Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality, China